CLINICAL TRIAL: NCT05574816
Title: Evaluation of the Diagnostic Performance of a Bra Prototype to Detect Breast Cancer
Acronym: Phi-Bra
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 69HCL21_1085
Record Dates: First submitted 2022-10-07; First posted 2022-10-12 (Actual); Last update posted 2024-06-12 (Actual); Status verified 2024-06

CONDITIONS: Breast Neoplasm Female
Keywords: Breast cancer detection; impedance

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Patient without breast lump (Active Comparator): No breast lump identified during mammography (ACR 1 et 2 Birads classification)
  Interventions: Device: Phi-Bra prototype measurements
- Patient with breast lump (Experimental): Suspicious breast lump identified during mammography (ACR 4b, c ou ACR 5 Birads classification)
  Interventions: Device: Phi-Bra prototype measurements

INTERVENTIONS:
Device: Phi-Bra prototype measurements — The bra prototype will be placed on the patient's breast. The patient will stay in a half-lying position during 15 min, the time duration of the measurements. Measurements will not be painful.
  Measurements will only be realized one time during the first and unique visit of the patient.

SUMMARY:
Phi-Bra is a prospective and monocentric pilot study to assess the diagnostic capability of an innovative bra prototype to detect breast cancer, compared to the current standard of care: the mammography.

The Phi-Bra prototype is designed with sensors measuring different parameters simultaneously such as impedance and temperature.

The bra will be tested on patients without breast lump (American College of Radiology (ACR) 1 et 2 Birads classification) and with breast lump (ACR 4b, c ou ACR 5 Birads classification).

The aim of this pilot study is to compare the results obtained by Phi-Bra to the ones obtained by mammography.

The Phi-Bra study is classified as clinical investigation category 4.4 based on the European Union (EU) regulation (DM 2017/745).

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 75.
* No breast cancer surgery background
* Bra size : S/M or M/L

Specific criteria for the "no breast lump" cohort:

- Negative mammography result (ACR 1 a 2).

Specific criteria for the "breast lump" cohort:

- Suspicious breast lump discovered during the mammography (ACR 4b ou c ou ACR 5) and for which there is an indication of microbiopsy.

Exclusion Criteria:

* Breast cancer background (surgery or radiotherapy)
* Breast lump classified as ACR 3 ou ACR 4a during the mammography

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2023-03-30 (Actual); Primary Completion 2024-02-01 (Actual); Study Completion 2024-02-01 (Actual)

PRIMARY OUTCOMES:
Aria Under Receiver Operating Characteristic (ROC) Curve | The day of inclusion
  The diagnostic performance of Phi-Bra to assess breast lump will be assessed by evaluating the ROC Area Under Curve (AUC), the reference being mammography as gold standard.

SECONDARY OUTCOMES:
impedance optimal threshold | The day of inclusion
  Determination of the impedance optimal threshold to detect breast lump in term of specificity and sensitivity (in Ohms)
Correlation between lump volume and device impedance | The day of inclusion

CONTACTS AND LOCATIONS:
Overall Officials: Marion CORTET, MD, PhD, Principal Investigator — Hospices Civils de Lyon
Locations (2):
- France (2):
  - Service de Gynecologie-Obstetrique, Hopital de la Croix Rousse, Lyon
  - Service de Radiologie, Hôpital de la Croix-Rousse, Lyon

IPD SHARING:
Plan to Share IPD: No